CLINICAL TRIAL: NCT01965587
Title: RCT Novasure Versus Novasure + Mirena IUS in the Treatment of Menorrhagia. A Pilot Study
Brief Title: RCT Novasure Versus Novasure + Mirena IUS in the Treatment of Menorrhagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Walsall Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Mr jonathan pepper MD FRCOG, Consultant Gynaecologist, Walsall Healthcare NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Novasure2013
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Menorrhagia
Keywords: novasure; Mirena IUS; menorrhagia; pelvic pain; ashermanns
MeSH Terms: conditions — Menorrhagia; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- novasure mirena IUS combined (Active Comparator): novasure mirena IUS combined therapy
  Interventions: Procedure: novasure mirena IUS combined
- novasure alone (Active Comparator): Sole treatment with Novasure
  Interventions: Procedure: novasure mirena IUS combined

INTERVENTIONS:
Procedure: novasure mirena IUS combined — novasure mirena IUS combined
  Other Names: Combined treatment Novasure and Mirena IUS

SUMMARY:
Hypothesis. Combined treatment with novasure and mirena IUS confers benefit over Novasure alone in the treatment of menorrhagia

DETAILED DESCRIPTION:
Endometrial ablation is a commonly used treatment option for women with heavy periods. It is recommended as an initial treatment. It aims at destroying the lining of the womb to reduce heavy menstrual loss.

A hormone releasing device in the womb (MIRENA®)is another commonly used treatment for women with heavy menstrual bleeding and has added benefit of reducing cyclical pain.

There is an increase in the number of women presenting to gynaecology clinic with persistence of pain or cyclical pain with absent or light bleeding after second generation endometrial ablation (Novasure). This may be due to the pockets of active lining of the womb that remains after ablation or possible adhesions created by the treatment. Most women require surgical removal of the womb (hysterectomy) because of pain or a further surgical procedure to divide these adhesions in an attempt to relieve pain and drain any collections in the womb.

We aim to determine if the combined use of MIRENA® and NOVASURE® (which is the second generation endometrial ablation technique used in our unit) will help in reducing the number of women presenting with cyclical pain and requiring further intervention or surgery. The aim of the current study is to compare between women receiving only NOVASURE treatment and women receiving combined NOVASURE and MIRENA treatment for heavy menstrual bleeding. The primary and secondary outcomes will be assessed at 6 and 12 months by a patient questionnaire. The primary outcome is improvement in quality of life The secondary outcomes include

* Lowering of surgical intervention
* Reduction in pain
* Reduction in amount of bleeding This will be a pilot study to determine if the theory is correct and then a larger powered study can be undertaken

ELIGIBILITY:
Inclusion Criteria:

* Anybody suitable for novasure ablation

Exclusion Criteria:

* Mirena IUS is indicated as treatment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 6 months
  Patient questionaire to assess periods and pain

CONTACTS AND LOCATIONS:
Locations (1):
- Walsall Manor Hospital, Walsall, West Midlands, United Kingdom